CLINICAL TRIAL: NCT04906330
Title: Oncoliq: Test for Early Breast Cancer Detection.
Status: Recruiting | Type: Observational
Sponsor: Hospital Militar Central Cirujano Mayor Dr. Cosme Argerich (Other)
Collaborators: Instituto Nacional del Cáncer, Argentina (Other Government)
Responsible Party: Principal Investigator, Adriana De Siervi, Ph.D.; Principal Investigator, Hospital Militar Central Cirujano Mayor Dr. Cosme Argerich
Other Study IDs: V1 11.12. 2020 (C.I.R.E.C.); IS003208 (Registry Identifier: RENIS)
Record Dates: First submitted 2021-05-13; First posted 2021-05-28 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Breast Cancer
Keywords: Liquid biopsy, breast cancer, early detection, microRNAs.
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — The plasma from participants will be obtained by centrifugation of blood collected with EDTA, and retained in a -80 ° C freezer exclusively for laboratory use and under lock and key. Samples will be codified and labelled.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- PPHM-0000-21: 50-70 year old female patients, without a personal history of oncological pathology, who attend for gynecological and mammographic control.
  Interventions: Diagnostic Test: Oncoliq: test for early breast cancer detection.

INTERVENTIONS:
Diagnostic Test: Oncoliq: test for early breast cancer detection. — Oncoliq is a novel early detection breast cancer test based on liquid biopsies and miRNAs. The main advantage of this test is that miRNAs released from the tumor into the bloodstream can be detected in the plasma of patients even when the tumor is undetectable by other methods.

SUMMARY:
Oncoliq is a novel early breast cancer detection test based on liquid biopsies and microRNAs. This innovative test will allow improving the accuracy of cancer detection which will impact on health, reducing the patient mortality and health costs.

To develop this test, it has been finished the preclinical PHASE I: in laboratory animals; PHASE II: exploratory clinical phase for the discovery of candidate biomarkers in breast cancer patients and PHASE III: clinical validation of biomarkers showing that Oncoliq has 91% of sensitivity.

Currently it is been setting up a "pilot test" for breast cancer to enrol 500 woman volunteers without previous cancer diagnosis that go to the annual medical control. The results of the pilot test will give the accuracy for early breast cancer detection.

ELIGIBILITY:
Inclusion Criteria:

* Women patients performing gynecological control
* Between 50-70 years old
* Without personal history of oncological disease
* Informed consent signed

Exclusion Criteria:

* Patients who don´t meet the inclusion criteria.
* Active infection with SARS-CoV-2 (COVID-19).

Ages: 50 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Female patients, without a personal history of oncological pathology, who attend for gynecological and mammographic control.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2024-08-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
miRNA levels in plasma | Day 1
  miRNA levels in plasma will be determined by RT-qPCR.

CONTACTS AND LOCATIONS:
Overall Officials: Adriana De Siervi, PhD, Principal Investigator — IBYME-CONICET
Locations (1):
- Hospital Militar Central, CABA, Buenos Aires, Argentina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Notice in a local online newspaper — https://www.infobae.com/sociedad/2020/08/22/como-es-el-innovador-kit-argentino-que-promete-detectar-el-cancer-de-mama-y-el-de-prostata-antes-que-los-analisis-tradicionales/
- See also: Notice in a local TV-news program — https://youtu.be/MeSAcWYHiEU